CLINICAL TRIAL: NCT07108361
Title: "Osseodensification Efficacy on Molar Septum Expansion in Immediate Molar Implant Placement: A Randomized Controlled Clinical Trial
Brief Title: "Osseodensification Efficacy on Molar Septum Expansion in Immediate Molar Implant Placement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Augusta University (Other)
Responsible Party: Principal Investigator, Mohammed Samir, Assistant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-REC ID052505
Record Dates: First submitted 2025-07-08; First posted 2025-08-07 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Implant Osseointegration; Implant Osteotomy; Implant Placement; Implant Primary Stability; Molar Extraction Socket; Immediate Implant Placement
Keywords: non restorable tooth; molar extraction; multirooted teeth; extraction socket; immediate Implant placement; Osseodensification; ex-vivo; RCT; Jumping gap; Grafting

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional drilling group (Active Comparator)
  Interventions: Procedure: conventional drilling
- Osseodensification group (Experimental)
  Interventions: Procedure: Osseodensification

INTERVENTIONS:
Procedure: Osseodensification — Septum width will be directly measured post molar extraction confirming the premeasure of the CBCT. Measurement will be recorded at the narrowest width of the septum. Implant site preparation starts with a pilot drill, in clockwise motion, in the center of the septum, until 1 mm deeper than the planned implant length. Densah® Burs (Versah, LLC, Jackson, MI, USA) were then sequentially used in OD mode (counterclockwise, drilling speed 800-1500 rpm, with copious irrigation) in small increments to gradually expand the osteotomy, until reaching the desired width for the planned implant diameter, Osteotomy diameter as a reflection of septum width expansion will then be directly measured and recorded after site instrumentation. Implants of adequate diameter (4, 4.5, or 5mm) and length (selected using preoperative CBCT) will be inserted in the prepared osteotomies to engage the bone apical to the socket, insertion torque will be measured using the torque wrench and ISQ values
  Arms: Osseodensification group
Procedure: conventional drilling — Septum width will be directly measured post molar extraction confirming the premeasure of the CBCT. Measurement will be recorded at the narrowest width of the septum. The initial (pointed) drill will be used to make a hole (starting point) in the interradicular bone to avoid slippage of the subsequent the drills in the socket of the remaining roots. The drills of increasing diameters will be used to complete the implant osteotomy according to manufacturer instructions. In case of limited interradicular bone volume, drilling will be made at the socket of mesial or distal roots. Osteotomy diameter as a reflection of septum width expansion will then be directly measured and recorded after site instrumentation. Implants of adequate diameter (4, 4.5, or 5mm) and length (selected using preoperative CBCT) will be inserted in the prepared osteotomies to engage the bone apical to the socket insertion torque will be measured using the torque wrench and ISQ values
  Arms: conventional drilling group

SUMMARY:
The ideal positioning of immediate implants in molar extraction sockets often requires the osteotomy to be in the interradicular septum, which can be challenging in some cases, with traditional site preparation techniques. Also, the alveolar ridge undergoes various remodeling processes following tooth extraction, resulting in hard and soft tissue loss which complicates prosthodontic rehabilitation. Immediate implant placement help preserve the alveolar ridge dimensions and buccal ridge contour. While osseodensification has shown promise in enhancing primary stability and bone microarchitecture, its clinical and microstructural effects in molar extraction sockets remain underexplored. Although there is ample documentation of information on the temperature that is generated during preparation of implant sites, there are no studies available in the literature comparing conventional drilling and osseodensification techniques; therefore, the present investigation was aimed at analyzing the efficacy of osseodensification compared to conventional drilling in terms of bone dimensions preservation , changes in bone architecture during implant site preparation and heat generation to define which technique can be safely applied to achieve the necessary implant primary stability without damaging the surrounding bone.

Aim of the study:

Is to compare the molar septum dimensions using osseodensification expansion versus the conventional drilling protocol and to assess the role of jumping gap grafting in preservation of the alveolar ridge dimensions and buccal ridge contour in addition to Evaluation of the effect of osseodensification on the bony micro-architecture and heat generation

DETAILED DESCRIPTION:
The proposed study consists of two arms: 1- Clinical arm, 2- Ex-Vivo arm

The clinical arm:

80 patients with hopeless teeth requiring extraction in the molar region and requiring replacement with dental implants, will be enrolled and recruited from the outpatient clinic, faculty of dentistry, Ain shams university according to the inclusion criteria. They will be randomly allocated into two equal groups. 40 patients in the osseodensification group and 40 patients in the conventional drilling group. Each group will be further subdivided into two groups with and without jumping gap graftingPerioperative and postoperative CBCT will be ordered, and perioperative and postoperative impressions will be made and scanned for each patient to prepare a virtual 3D model before extraction and after extraction and implant placement. Molar septum dimensions will be compared before and after implant placement in addition to evaluation of vertical and horizontal alveolar bone changes and changes in bone density after placement of immediate implant in extraction socket, also a volumetric analysis will be made to assess the changes in the buccal ridge contour before and after implant placement with and without grafting of the jumping gap. Clinical outcomes will be assessed including (success and survival of implants, insertion torque, ISQ values, Probing depth, modified pink esthetic score, KTW, and patient satisfaction) all the outcomes will be assessed as baseline before the implant placement and will be followed up at 0,6 and 12 months after implant placementThe Ex-Vivo arm: study will be conducted in an ex vivo animal model using porcine bones. The animals won't be used exclusively for this study and the bones will be collected as if it was disposable as waste material, so ethical approval will not be necessary. Both tibias of a single skeletally mature porcine will be collected on the day of the slaughter. To prepare the samples, approximately 15 mm of the articular surface and subchondral bone will be removed by transversely sectioning the bones, thereby exposing the medullary portion. Three canals for thermocouples at three different depths (2 mm: T1-cortical bone, 7.5 mm: T2-cancellous bone, and 10.5 mm: T3- deep cancellous bone) from the crest of the pig bone will be drilled using 1.5 mm twist drill perpendicularly to each implant site preparation and using intermittent cutting to a distance approximately 1 mm from the planned osteotomy site.The thermocouples will be secured to the bone blocks at a distance of approximately 1 mm from the future osteotomy and insulated using sticky wax at the canal opening This study will be performed on 12 samples removed from the tibias, divided into two groups according to the drilling technique: a control group of the conventional technique (CT) (n=6), and a test group of osseodensification (OD) (n=6). The evaluation of bone microstructure using Micro-CT will follow the guidelines proposed by Bouxsein et al. (2010), which includes the use of terminologies, procedures, images, and reporting of the results. The thermocouples will be connected to a digital thermometer that allows continuous temperature reading, and temperature changes (baseline and final temperature readings) during the osteotomy preparation will be recorded for statistical analysis

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring placement in the posterior region.

  * ASA I and II patients who can undergo immediate implant placement and restorative procedures.
  * Both males and females.
  * Patient's age: 18-50 years old.
  * Patients who can come for the follow-up visit.
  * Patients who provide written informed consent

Exclusion Criteria:

* Pregnancy.

  * Smoking
  * Patients with previously failed dental implants at the implant placement site.
  * Patients with active infections.
  * Other medical conditions that might affect the osseointegration of dental implants, such as diabetes, cardiovascular disease, hypertension, and osteoporosis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment of molar septum dimensional changes of the extraction socket following osseodensification and conventional drilling protocols | from enrollment to the day of surgery
  Septum width will be directly measured post molar extraction. Measurement will be recorded at the narrowest width of the septum Osteotomy diameter as a reflection of septum width expansion will then be directly measured and recorded after site instrumentation

SECONDARY OUTCOMES:
Comparing of bony Micro-architecture following osseodensification and conventional drilling protocols. | Day of surgery
  Micro-CT imaging osteotomy sites bone samples will be performed using a SkyScan 1272 microfocus X-ray system (SkyScan®, Kontich, Belgium) with software including NRecon reconstruction®, CTAn 1.8®, and CTvol. In this study, the X-ray source will be set at 70 kV and 100μA with the pixel size of 6μm, a 0.5-mm filter, and a tomographic rotation of 180° (rotation step of 0.2°). Residual bone volume (BV, μm3) around osteotomy sites will be quantified and 3-D models will be generated
Comparing amount of heat generation following osseodensification and conventional drilling protocols. | from enrollment to the day of surgery
Assessment of the clinical outcomes of implant placement in the extraction socket comparing the two drilling protocols | All parameters will be assessed immediately after implant placement (T0), six months (T6) and 12 months (T12)
  Implant ISQ values
Radiographic assessment of molar septum dimensional changes of the extraction socket following osseodensification and conventional drilling protocols | All parameters will be assessed immediately after implant placement (T0), six months (T6) and 12 months (T12)
> Volumetric assessment of the ridge buccal contour following implant placement with and without grafting the jumping gap. | All parameters will be assessed preoperative, six months (T6) and 12 months (T12)
  comparing ridge volume changes before and after surgery with and without grafting
Evaluation of Patient satisfaction | day of surgery to 12 months after loading
  Te patient satisfaction for aesthetics, function, sense, speech, and self-esteem was evaluated by a numeric rating scale ranging from 0 to 5, where 0 represents "very dissatisfed" and 5 represents "very satisfed"
Radiographic assessment of the vertical and horizontal dimensional changes of the alveolar ridge following implant placement comparing the 2 drilling protocols and comparing the effect of jumping gap grafting | measurements will be performed on CBCT images taken immediately after implant placement (T0), six months (T6) and 12 months (T12)
  Radiographic evaluation of vertical and horizontal alveolar bone changes will be performed on CBCT images taken immediately after implant placement (T0), six months (T6) and 12 months (T12). The following distances will be measured around the four implants surfaces; 1) P-BIC; from implant platform to the first bone contact, 2) P-T; vertical distance between implant platform and alveolar bone crest, 3) OBS; from buccal and lingual border of bone to the implant surface at the level of the implant platform (OBS0), 2 mm (OBS2), and 4 mm (OBS4) apical to implant platform.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No